CLINICAL TRIAL: NCT03429712
Title: Patient- and Task-specific Radiation Dose Optimization for Pediatric Abdominopelvic CT Applications
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to slow enrollment.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00077173
Record Dates: First submitted 2018-02-06; First posted 2018-02-12 (Actual); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Split Dose CT
Keywords: CT Scan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dose Split CT (Experimental)
  Interventions: Device: Dual-source multi-detector computed tomography (DSSE)

INTERVENTIONS:
Device: Dual-source multi-detector computed tomography (DSSE) — Dose split technique in a cohort of pediatric patients to determine, without increase in patient radiation dose, the optimal patient-specific and task-specific radiation dose levels for pediatric cardiothoracic and abdominal CT applications.

SUMMARY:
Radiation dose reduction has been a primary driver of technology development in multi-detector computed tomography (MDCT). The optimization of radiation dose for patient and task specific computed tomography (CT) applications continues to be an ongoing challenge, especially in pediatric patients where the desire to reduce radiation dose to lowest possible levels leads to both positive and negative effects. A novel research tool on the Siemens dual source (Flash® and Force ®) CT scanners allows one to assess multiple tube current levels from a single CT acquisition without incurring additional dose to the patient. Tube current is a primary contributor to radiation dose and image noise, which are inversely related. This is achieved by independently adjusting the current of each tube, while maintaining same kV in each x-ray tube. Moreover, Duke's medical physics team has developed a method based on mathematical expressions that allows the creation of incremental dose levels from the acquired image data sets. This innovative and powerful tool can be used to compare diagnostic accuracy, detectability, and many more relevant clinical features amongst multiple tube current levels with the attainment of a single CT acquisition.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Pregnant

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Marin, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Split CT
Started | 19
Completed | 10
Not Completed | 9

BASELINE CHARACTERISTICS:
Population: Subjects who completed the study.
Arm/Group | Dose Split CT
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.56 (5.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Image Noise
Time Frame: Up to 5 minutes
Population: Data not collected.
Arm/Group | Dose Split CT
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: The patients were at very low risk for serious adverse events, mortality, or any other adverse event due to the different methodology used to deliver the same radiation dose the patient would have received in a standard abdomen and pelvis CT.
Arm/Group | Dose Split CT
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT03429712/Prot_SAP_000.pdf